CLINICAL TRIAL: NCT04727892
Title: Severity Grading, Risk Factors and Prediction Model of Complications After Epilepsy Surgery: a Single-center, Large-scale and Retrospective Study
Brief Title: Complications After Epilepsy Surgery
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Zhang Hua, Doctor, First Affiliated Hospital Xi'an Jiaotong University
Other Study IDs: XJTU1AF2020LSK-167
Record Dates: First submitted 2021-01-18; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Epilepsy; Surgery--Complications
Keywords: epilepsy surgery; complication; prediction
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- complications after epilepsy surgery: Group A with no complication; Group B with complications
  Interventions: Procedure: epilepsy surgery

INTERVENTIONS:
Procedure: epilepsy surgery — Surgical procedures were individually designed according to the presurgical evaluation findings. Standard epilepsy surgery procedures were applied. Generally, surgical procedures were divided into curative and palliative surgery. Curative surgery included resection and disconnection of the epileptogenic zone. Palliative surgery included corpus callosotomy for bilateral synchronous onset and multiple subpial transections for epileptic foci located in the eloquent cortex. For widespread epileptogenic zones, multiple surgical techniques were combined.

SUMMARY:
Epilepsy surgery is effective for refractory epilepsy, particularly focal epilepsy, but is still underutilized worldwide. In the United States, the annual percentage of surgical procedures for refractory epilepsy was low (range: 0.35%-0.63%) from 2003 to 2012. Fear associated with the risks of invasive procedures may be the reason for the cautious attitude towards epilepsy surgery. Therefore, the risks of epilepsy surgery in the modern age need to be evaluated thoroughly and precisely to improve epilepsy surgery outcomes.

The safety of epilepsy surgery has been confirmed in several studies. Studies on this topic with large sample sizes (> 500 patients) were either multicenter or covered a long study period. In addition, high-resolution magnetic resonance imaging (MRI) was not used in the early stage in these studies. Differences in medical environment among epilepsy centers and advancements in presurgical evaluations and surgical techniques over time may have caused heterogeneity and biases, thereby limiting the quality of these studies. Over the past two decades, there was no large-scale studies on post-epilepsy surgery complications performed at a single center. Moreover, surgery-related complications are seldom graded according to severity. Especially, the risk factors for these complications remain unclear.

DETAILED DESCRIPTION:
Epilepsy, involving a persistent predisposition to seizure, is one of the most common chronic neurological disorders, affecting more than 65million people worldwide. Epilepsy not only negatively impacts patients'education, employment, and social contact, but also imposes a serious burden on patients'families and on society. Notably, epilepsy is the second most burdensome neurological disorder, accounting for 0.7% of disability-adjusted life years worldwide, according to the World Health Organization's 2010 Global Burden of Disease study, making it a global public health issue.

Furthermore, about 40% of patients respond poorly to the first 2 antiepileptic drugs and have medically refractory epilepsy. Epilepsy surgery is effective for refractory epilepsy, particularly focal epilepsy, but is still underutilized worldwide. In the United States, the annual percentage of surgical procedures for refractory epilepsy was low (range: 0.35%-0.63%) from 2003 to 2012. Moreover, the number of surgical procedures for mesial temporal sclerosis (the most common type of refractory epilepsy) declined by more than half from 2006 to 2010. Fear associated with the risks of invasive procedures may be the reason for the cautious attitude towards epilepsy surgery. Therefore, the risks of epilepsy surgery in the modern age need to be evaluated thoroughly and precisely to improve epilepsy surgery outcomes.

The safety of epilepsy surgery has been confirmed in several studies. From 1980 to 2012, neurological deficits following epilepsy surgery decreased with time, from 41.8% to 5.2% in temporal resections and from 30.2% to 19.5% in extratemporal resections. However, studies on this topic with large sample sizes (> 500 patients) were either multicenter or covered a long study period. In addition, high-resolution magnetic resonance imaging (MRI) was not used in the early stage in these studies. Differences in medical environment among epilepsy centers and advancements in presurgical evaluations and surgical techniques over time may have caused heterogeneity and biases, thereby limiting the quality of these studies. Over the past two decades, there was no large-scale studies on post-epilepsy surgery complications performed at a single center. Moreover, surgery-related complications are seldom graded according to severity. Especially, the risk factors for these complications remain unclear.

Understanding the incidence and severity of complications after epilepsy surgery and the associated risk factors is beneficial, allowing physicians to provide patients with adequate surgical advice, and allowing patients to make rational decisions regarding epilepsy surgery. Furthermore, this information may help in the prevention of postoperative complications and improve our understanding of the procedures. Therefore, we reported the incidence of complications occurring in a three-month period after epilepsy surgery performed by the single neurosurgeon at the single center, identified the associated risk factors, and developed a nomogram for individually predicting the probability of complications.

ELIGIBILITY:
Inclusion Criteria:

* (i) medically refractory epilepsy defined by the International League Against Epilepsyc; (ii) epilepsy surgery performed by a single neurosurgeon, Dr. H.Z.; (iii) surgical procedure performed via craniotomy.

Exclusion Criteria:

* Patients with neuromodulation therapy were excluded in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a large-scale retrospective study of patients undergoing epilepsy surgery performed by a single neurosurgeon, Dr. Zhang, at the single epilepsy centre from.
Sampling Method: Non-Probability Sample
Enrollment: 2026 (Actual)
Dates: Start 2003-10-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Complications | in the 3-month period after epilepsy surgery
  Complications included neurologic deficit, cerebral edema, intracranial hemorrhage, infection, hydrocephalus, subdural effusion, subcutaneous cerebrospinal fluid accumulation, and poor wound healing. Neurologic deficit was classified as either transient (resolving within 3 months) or persistent (lasting more than 3 months) Complication severity was categorized into four grades based on the therapeutic regimen: grade I, minor complications, conservative treatment; grade II, major complications; grade III, life-threatening complications requiring invasive treatment under general anesthesia or monitoring in the intensive care unit; grade IV, death.

SECONDARY OUTCOMES:
Predictors of complications. | in the 3-month period after epilepsy surgery
  Potential factors included the preoperative, intra-operative, and postoperative clinical characteristics, such as sex, age at surgery, duration of seizure, previous medical history, pathology, serial number of surgery, invasive electrode implantation, type of surgical procedure, surgery duration, intra-operative blood loss, and acute postoperative seizure.
  Risk factors for complications were determined by using univariate and multivariate logistic regression analyses. Variables with P< .10 were selected as a potential risk factors and included in the multivariate logistic regression analysis. The forward stepwise method was used to select the variables that were eventually included in the model. Odds ratio (OR) and 95% confidence interval (CI) were calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Zhang, PhD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University

IPD SHARING:
Plan to Share IPD: Yes
Partial participant data are to be shared with other researchers
Supporting Information: SAP, CSR
Time Frame: 0ct 2021, for 1 month
Access Criteria: clinical study